CLINICAL TRIAL: NCT00978380
Title: A Multi-Centre, Open-Label, Single-Arm, and Multiple Dosing Trial on Safety of Monthly Replacement Therapy With Recombinant Factor XIII (rFXIII) in Subjects With Congenital Factor XIII Deficiency
Brief Title: Safety of Monthly Recombinant Factor XIII Replacement Therapy in Subjects With Congenital Factor XIII Deficiency: An Extension to Trial F13CD-1725
Acronym: mentor™2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: F13CD-3720; 2008-007883-41 (EudraCT Number); U1111-1111-9289 (Other: WHO); JapicCTI-121958 (Registry Identifier: JAPIC)
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Results first posted 2016-12-13 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Congenital Bleeding Disorder; Congenital FXIII Deficiency
MeSH Terms: interventions — recombinant factor XIII-A2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: catridecacog

INTERVENTIONS:
Drug: catridecacog — Monthly administration of recombinant factor XIII as preventative treatment of bleeding episodes. Dose: 35 IU/kg body weight intravenous (into the vein)
  Other Names: recombinant factor XIII

SUMMARY:
This trial is conducted in Asia, Europe and North America. The aim of the trial is to investigate the safety of monthly replacement therapy of recombinant factor XIII in patients with congenital FXIII deficiency. The trial continues until the product is commercially available, but an interim assessment will take place when all subjects have completed 52 weeks in the trial.

ELIGIBILITY:
Inclusion Criteria:

* For subjects who participated in F13CD-1725:
* Previous participation (means up to and inclusive Visit 16, (End of Trial)) in F13CD-1725
* For all other subjects:
* Diagnosis of congenital FXIII A-subunit deficiency (confirmed by genotyping at screening visit or documented results from previously performed genotyping)
* Body weight at least 20 kg

Exclusion Criteria:

* Known neutralizing antibodies (inhibitors) towards FXIII
* Any known congenital or acquired coagulation disorder other than congenital FXIII deficiency
* Platelet count (thrombocytes) of less than 50 × 109/L. For subjects who participated in F13CD-1725 platelet count from visit 15 in F13CD-1725 must be used for evaluation.
* Females of childbearing potential who are pregnant, breastfeeding or are not using adequate contraceptive methods

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2009-09-21 (Actual); Primary Completion 2015-10-20 (Actual); Study Completion 2015-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (34):
- United States (12):
  - Novo Nordisk Investigational Site, Orange, California
  - Novo Nordisk Investigational Site, Washington D.C., District of Columbia
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Boise, Idaho
  - Novo Nordisk Investigational Site, Detroit, Michigan
  - Novo Nordisk Investigational Site, Minneapolis, Minnesota
  - Novo Nordisk Investigational Site, Columbus, Ohio
  - Novo Nordisk Investigational Site, Oklahoma City, Oklahoma
  - Novo Nordisk Investigational Site, Hershey, Pennsylvania
  - Novo Nordisk Investigational Site, Richmond, Virginia
  - Novo Nordisk Investigational Site, Seattle, Washington
- Novo Nordisk Investigational Site, Klagenfurt, Austria
- Novo Nordisk Investigational Site, Toronto, Ontario, Canada
- Novo Nordisk Investigational Site, Helsinki, Finland
- France (4):
  - Novo Nordisk Investigational Site, Le Kremlin-Bicêtre
  - Novo Nordisk Investigational Site, Paris
  - Novo Nordisk Investigational Site, Rouen
  - Novo Nordisk Investigational Site, Valence
- Germany (3):
  - Novo Nordisk Investigational Site, Bonn
  - Novo Nordisk Investigational Site, Braunschweig
  - Novo Nordisk Investigational Site, Duisburg
- Novo Nordisk Investigational Site, Petah Tikva, Israel
- Novo Nordisk Investigational Site, Vicenza, Italy
- Japan (2):
  - Novo Nordisk Investigational Site, Hiroshima-shi, Hiroshima
  - Novo Nordisk Investigational Site, Shinjuku-ku, Tokyo
- Spain (3):
  - Novo Nordisk Investigational Site, Barcelona
  - Novo Nordisk Investigational Site, Málaga
  - Novo Nordisk Investigational Site, Tortosa
- Novo Nordisk Investigational Site, Zurich, Switzerland
- United Kingdom (4):
  - Novo Nordisk Investigational Site, Aberdeen
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Manchester
  - Novo Nordisk Investigational Site, Newcastle upon Tyne

REFERENCES:
- [Result] Brand-Staufer B, Carcao M, Kerlin BA, Will A, Williams M, Tornoe CW, Sandberg Lundblad M, Nugent D. Pharmacokinetic characterization of recombinant factor XIII (FXIII)-A2 across age groups in patients with FXIII A-subunit congenital deficiency. Haemophilia. 2015 May;21(3):380-385. doi: 10.1111/hae.12616. Epub 2015 Jan 21. PMID 25643920
- [Result] Kerlin B, Brand B, Inbal A, Halimeh S, Nugent D, Lundblad M, Tehranchi R. Pharmacokinetics of recombinant factor XIII at steady state in patients with congenital factor XIII A-subunit deficiency. J Thromb Haemost. 2014 Dec;12(12):2038-43. doi: 10.1111/jth.12739. Epub 2014 Oct 25. PMID 25263390
- [Derived] Byrnes JR, Lee T, Sharaby S, Campbell RA, Dobson DA, Holle LA, Luo M, Kangro K, Homeister JW, Aleman MM, Luyendyk JP, Kerlin BA, Dumond JB, Wolberg AS. Reciprocal stabilization of coagulation factor XIII-A and -B subunits is a determinant of plasma FXIII concentration. Blood. 2024 Feb 1;143(5):444-455. doi: 10.1182/blood.2023022042. PMID 37883802
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 34 sites in 12 countries as follows: Austria: 1 site; Canada: 1 site; Finland: 1 site; France: 4 sites; Germany: 4 sites; Israel: 1 site; Italy: 1 site: Japan: 2 sites; Spain: 2 sites; Switzerland: 1 site; United Kingdom: 4 sites; United States: 12 sites.
Pre-assignment Details: Subjects who completed F13CD-1725 (CT.gov identifier: NCT00713648) end of trial visit were eligible to enroll in this trial. Also, new subjects diagnosed with congenital FXIII A-subunit deficiency (confirmed by genotyping at screening visit or documented results from previously performed genotyping) were enrolled to expand the safety population.
Groups:
- Recombinant Factor XIII (rFXIII): Subjects received 35 IU/kg bodyweight of rFXIII slow intravenous (i.v.) injection every 4 weeks (28 days±2 days) for a minimum period of 52 weeks until the end of trial visit. The dose was identical to the dose administered in the F13CD- 1725 trial. A total of 60 unique subjects were enrolled and exposed in the trial, but 3 of these subjects were later withdrawn and subsequently re-enrolled with new subject IDs, giving rise to a total of N=63 subjects. The unique subjects (N=60) were presented as full analysis set (FAS) while summarising adverse events to avoid double-counting.
Period: Overall Study
Arm/Group | Recombinant Factor XIII (rFXIII)
Started | 63
Completed | 44
Not Completed | 19
Not completed — Protocol Violation | 2
Not completed — Withdrawal criteria | 9
Not completed — Unclassified | 8

BASELINE CHARACTERISTICS:
Population: All subjects who received trial product were considered for baseline characteristics including 3 subjects who were re-enrolled with new subject IDs.
Arm/Group | Recombinant Factor XIII (rFXIII)
Number analyzed (Participants) | 63
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31 (16.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 52
  Unknown or Not Reported | 4
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 37
  More than one race | 0
  Unknown or Not Reported | 4
  Other | 6

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events (AEs)(Serious and Non-serious)
Description: An AE was defined as any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Trial AEs (serious) included any event such as death, life-threatening experience, in-subject hospitalisation, significant disability/ congential anomaly experienced from the trial product.
Time Frame: All AEs were collected and reported from screening (week 0) for a minimum period of 52 weeks or until the end of trial visit.
Population: The FAS included the 60 unique subjects exposed to trial product in this extension trial.
Measure: Number; unit: Events
Arm/Group | Recombinant Factor XIII (rFXIII)
Number analyzed (Participants) | 60
Events
  All adverse events | 920
  Serious adverse events | 19
  Non-serious adverse events | 901

2. Secondary Outcome: Antibody and Inhibitor Development
Description: All subjects who received rFXIII were monitored for anti-rFXIII antibodies and inhibitor development. Samples passed through 2 tiers of ELISA testing: an initial screen with a specific cut-off point (including ~5% false positives) and a second confirmatory assay for samples yielding a result above the screening cut-off point. If samples were confirmed as antibody positive in the confirmation assay, an inhibitor assay was also carried out to detect functional inhibitors. Percentage of subjects with antibody and inhibitor development were reported.
Time Frame: From week 0 to week 52
Population: The safety analysis set included all subjects exposed to trial product in this extension trial.
Measure: Number; unit: Percentage of subjects
Arm/Group | Recombinant Factor XIII (rFXIII)
Number analyzed (Participants) | 63
Percentage of subjects | 0

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) were collected and reported from screening (week 0) for a minimum period of 52 weeks or until the end of trial visit.
Description: The FAS was used for AEs. In the early stage of the trial, a contract manufacturing facility (Avecia) produced the drug. Later, Novo Nordisk took over production of the drug. Hence, AE data are presented seperately who received both rFXIII Avecia and Novo Nordisk. Subsequently, subjects were counted under both groups.
Groups:
- rFXIII Novo Nordisk: Subjects in this arm received identical dose of 35 IU/kg bodyweight of rFXIII slow intravenous (i.v.) administered every 4 weeks (28 days±2 days) until the end of trial for a minimum period of 52 weeks. In the early stage of the trial, a contract manufacturing facility (Avecia) produced the rFXIII drug substance (rFXIII Avecia) and subsequently, Novo Nordisk took over production of the rFXIII drug substance (rFXIII Novo Nordisk). Characterisation testing between the two products confirmed that rFXIII Novo Nordisk and rFXIII Avecia had identical structures, and similar physico-chemical properties. The AE data are presented seperately for rFXIII Novo Nordisk and rFXIII Avecia. However, subjects in this arm received rFXIII Novo Nordisk drug.
- rFXIII Avecia: Subjects in this arm received identical dose of 35 IU/kg bodyweight of rFXIII slow intravenous (i.v.) administered every 4 weeks (28 days±2 days) until the end of trial for a minimum period of 52 weeks. In the early stage of the trial, a contract manufacturing facility (Avecia) produced the rFXIII drug substance (rFXIII Avecia) and subsequently, Novo Nordisk took over production of the rFXIII drug substance (rFXIII Novo Nordisk). Characterisation testing between the two products confirmed that rFXIII Novo Nordisk and rFXIII Avecia had identical structures, and similar physico-chemical properties. The AE data are presented seperately for rFXIII Novo Nordisk and rFXIII Avecia. However, subjects in this arm received rFXIII Avecia drug.
Arm/Group | rFXIII Novo Nordisk | rFXIII Avecia
Serious Adverse Events (participants affected / at risk) | 12/59 | 0/26
Other Adverse Events (participants affected / at risk) | 54/59 | 15/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rFXIII Novo Nordisk (N=59) | rFXIII Avecia (N=26)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Otitis media chronic (Infections and infestations) | 1 (1) | 0 (0)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Spinal cord injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rFXIII Novo Nordisk (N=59) | rFXIII Avecia (N=26)
Abdominal pain (Gastrointestinal disorders) | 5 (6) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 4 (6) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (24) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (12) | 2 (2)
Constipation (Gastrointestinal disorders) | 5 (5) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 11 (18) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (29) | 0 (0)
Dental caries (Gastrointestinal disorders) | 3 (4) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 6 (14) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 4 (4) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 8 (10) | 1 (1)
Fatigue (General disorders) | 3 (3) | 0 (0)
Folliculitis (Infections and infestations) | 3 (4) | 0 (0)
Gastroenteritis (Infections and infestations) | 8 (10) | 0 (0)
Haematuria (Renal and urinary disorders) | 3 (3) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 3 (4) | 1 (1)
Headache (Nervous system disorders) | 19 (72) | 2 (4)
Hypertension (Vascular disorders) | 3 (4) | 0 (0)
Incorrect dose administered (Injury, poisoning and procedural complications) | 6 (9) | 1 (1)
Influenza (Infections and infestations) | 7 (8) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 4 (6) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 6 (9) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 5 (8) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (5) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 (20) | 0 (0)
Nasopharyngitis (Infections and infestations) | 19 (48) | 2 (2)
Nausea (Gastrointestinal disorders) | 7 (8) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 (31) | 0 (0)
Pain (General disorders) | 3 (4) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (32) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 3 (4) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (5) | 0 (0)
Pyrexia (General disorders) | 6 (11) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 5 (8) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Seasonal allergy (Immune system disorders) | 3 (4) | 0 (0)
Sinusitis (Infections and infestations) | 11 (17) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 3 (4) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 6 (6) | 2 (2)
Tonsillitis (Infections and infestations) | 5 (8) | 0 (0)
Toothache (Gastrointestinal disorders) | 4 (6) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 14 (25) | 0 (0)
Viral infection (Infections and infestations) | 3 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 0 (0)
White blood cells urine positive (Investigations) | 3 (3) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)

LIMITATIONS AND CAVEATS:
Limitations of the trial include small number of children and adolescents (16 subjects), and the sensitivity of the Berichrome® FXIII activity assay. However, mean FXIII activity levels were consistent with few bleeds requiring haemostatic treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publication will be prepared collaboratively between Investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.